CLINICAL TRIAL: NCT03350230
Title: Embryonic Ploidy Status in the Oncofertility Population
Status: Completed | Type: Observational
Sponsor: Reproductive Medicine Associates of New Jersey (Other)
Responsible Party: Sponsor
Other Study IDs: RMA-2017-05
Record Dates: First submitted 2017-11-13; First posted 2017-11-22 (Actual); Last update posted 2023-05-03 (Actual); Status verified 2023-05

CONDITIONS: Oncology; Fertility
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood specimens and buccal swabs
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- oncofertility patients: oncofertility patients undering controlled ovarian hyperstimulation and embryo cryopreservation who carry a present or past cancer diagnosis

SUMMARY:
looking at aneuploidy rates in embryos from patients who are going to or have undergone treatment for a malignancy with gonadotoxic treatment.

DETAILED DESCRIPTION:
The study involves oncofertility patients--individuals who are undergoing or have undergone therapy for a malignancy--who are interested in pursuing or preserving fertility. In particular, it investigates chromosomal abnormalities or aneuploidy in the embryos of those individuals as compared to the general infertility population. Embryonic aneuploidy is largely due to reproductive senescence. As such the investigators will discuss oncofertility prevalence and treatment as well as reproductive senescence and assessment of embryonic aneuploidy. The study will seek to determine if there are changes in embryonic aneuploidy rates in oncofertility patients that differ from simple age related risks.

ELIGIBILITY:
Inclusion Criteria:

1.Present or past oncologic diagnosis requiring potentially gonadotoxic treatment

Exclusion Criteria:

1. Oocyte banking
2. Use of oocyte donation
3. Any contraindications to undergoing in vitro fertilization or gonadotropin stimulation
4. Single gene disorder requiring more detailed embryo genetic analysis

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: oncofertility patient undergoing controlled ovarian hyperstimulation and embryo cryopreservation
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2017-12-01 (Actual); Primary Completion 2020-03-27 (Actual); Study Completion 2022-07-21 (Actual)

PRIMARY OUTCOMES:
embryonic aneuploidy rates | 1 month
  to evaluate the incidence of embryonic aneuploidy among oncofertility patients compared to the general infertility population

CONTACTS AND LOCATIONS:
Overall Officials: Jason Franasiak, MD, Principal Investigator — Reproductive Medicine Associates of New Jersey
Locations (1):
- Reproductive Medicine Associates of New Jersey, Basking Ridge, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No